CLINICAL TRIAL: NCT01414075
Title: A Phase 2, Randomized, Open-Label, Dose Titration, Safety and Efficacy Study of FG-4592 for the Correction of Anemia in Newly Initiated Dialysis Patients Not on Erythropoiesis-Stimulating Agent Treatment
Brief Title: Study of Roxadustat (FG-4592) to Correct Anemia in Newly Initiated Dialysis Participants Not on Erythropoiesis-Stimulating Agent Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-053
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Results first posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Dialysis; Anemia
Keywords: Kidney; ESRD; Renal; End-Stage Renal Disease; Anemia; Oral anemia treatment; Hemoglobin levels; Hemodialysis; Peritoneal; HD; PD; Hb; Erythropoietin; Blood count
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic | interventions — roxadustat; Iron; ferryl iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A + E (Participants on HD): Roxadustat Only, No Iron (Experimental): Participants on HD will receive roxadustat capsules at the applicable dose (up to a maximum roxadustat dose of 140, 200, and 300 mg) based on weight and Hb level, administered orally 3 times weekly (TIW) for 12 weeks.
  Interventions: Drug: Roxadustat
- Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg (Experimental): Participants on HD will receive roxadustat capsules at the applicable dose (up to a maximum roxadustat dose of 140, 200, and 300 mg) based on weight and Hb level, administered orally TIW with iron (ferrous fumarate or ferrous gluconate) PO at doses containing elemental iron between 50 and 195 mg daily (depending on the type of iron formulation available in their countries) for 12 weeks.
  Interventions: Drug: Roxadustat; Drug: Oral Iron
- Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg (Experimental): Participants on HD will receive roxadustat capsules at the applicable dose (up to a maximum roxadustat dose of 140, 200, and 300 mg) based on weight and Hb level, administered orally TIW with approximately 60 mg IV iron (ferric gluconate complex in sucrose injection [for example, Ferrlecit®] or equivalent) once a week for 12 weeks.
  Interventions: Drug: Roxadustat; Drug: IV Iron
- Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg (Experimental): Participants on PD will receive roxadustat capsules at the applicable dose (up to a maximum roxadustat dose of 140, 200, and 300 mg) based on weight and Hb level, administered orally TIW with iron (ferrous fumarate or ferrous gluconate) PO at doses containing elemental iron between 50 and 195 mg daily (depending on the type of iron formulation available in their countries) for 12 weeks.
  Interventions: Drug: Roxadustat; Drug: Oral Iron

INTERVENTIONS:
Drug: Roxadustat — Tiered, weight-based dosing per schedule specified in the arm.
  Other Names: FG-4592
Drug: Oral Iron — Administered per oral dose and schedule specified in the arm.
  Arms: Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg; Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Drug: IV Iron — Administered per IV dose and schedule specified in the arm.
  Arms: Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of roxadustat in the correction of anemia in participants with end-stage renal disease who recently started dialysis.

DETAILED DESCRIPTION:
Participants on hemodialysis (HD) will be randomized to 3 treatment arms (A, B, and C) of in a 1:1:1 ratio to receive no iron supplementation, oral iron supplementation, and IV iron supplementation, respectively, in addition to roxadustat. At the same time, participants on peritoneal dialysis (PD) will be enrolled into Arm D. Arm E will enroll either HD or PD participants, and is an optional, confirmatory/supplemental treatment arm with flexible dosing and flexible iron supplementation based on the evaluation of data from the previous 4 treatment arms.

Initial roxadustat dose will be based on a tiered, weight-based dosing scheme (low weight [40 to 60 kilograms {kg}], medium weight [>60 to 90 kg], and heavy weight [>90 to 140 kg] participants will receive 60, 100, and 140 milligrams [mg] roxadustat, respectively). Dose adjustments will be implemented (up to a maximum roxadustat dose of 140, 200, and 300 mg for low, medium, and high weight participants, respectively) during Weeks 5 and 9, depending on the hemoglobin (Hb) level and rate of Hb rise in the previous 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Receiving HD or PD for native kidney end-stage renal disease (ESRD) for 2 weeks to 4 months, prior to randomization
* Mean of the 2 most recent Hb values during the screening period, obtained at least 7 days apart, must be <10.0 grams (g)/deciliter (dL), with a difference of ≤1.0 g/dL between the 2 values
* Body weight 40 to 140 kilograms (kg)

Exclusion Criteria:

* Previously received erythropoiesis-stimulating agents
* Received IV iron within 4 weeks of randomization
* Received red blood cell transfusion within 8 weeks prior to randomization or anticipated need for transfusion during the treatment period
* Positive for any of the following: human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus antibody (anti-HCV Ab)
* History of chronic liver disease
* Clinically significant infection
* New York Heart Association Class III or IV congestive heart failure
* History of malignancy, except the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps
* Chronic inflammatory disease that could impact erythropoiesis (for example, systemic lupus erythematosis, rheumatoid arthritis, celiac disease) even if it is currently in remission
* History of other blood disorders
* Active hemolysis or diagnosis of hemolytic syndrome
* Known bone marrow fibrosis
* Uncontrolled or symptomatic secondary hyperparathyroidism
* History of alcohol or drug abuse within a year prior to randomization, or anticipated inability to avoid consumption of more than 3 alcoholic beverages per day
* History of allergy or sensitivity to oral or IV iron therapy
* Seizure disorder or receiving anti-epilepsy medication for seizure disorder within 12 weeks prior to randomization
* Pregnant or breast-feeding females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07-21 (Actual); Primary Completion 2013-01-10 (Actual); Study Completion 2013-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Northridge, California
  - Yuba City, California
  - Detroit, Michigan
- Hong Kong, Hong Kong
- Russia (2):
  - Moscow
  - Saint Petersburg
- Singapore, Singapore

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants on hemodialysis (HD) were randomized to one of the 3 arms A, B, or C in 1:1:1 ratio to receive roxadustat with either no, per oral (PO), or intravenous (IV) iron supplementation, respectively. Participants on peritoneal dialysis (PD) were enrolled into Arm D and received roxadustat with PO iron supplementation.
Pre-assignment Details: Arm E was an optional, confirmatory/supplemental arm with flexible dosing and flexible iron supplementation based on the evaluation of data from the previous 4 arms. After enrollment of Arms A through C was completed, Arm E was decided to be identical to Arm A, for example, roxadustat with no iron supplementation and with the same tiered weight-based initial dosing. Hence, the data of Arms A and E were reported in a single arm.
Groups:
- Arm A + E (Participants on HD): Roxadustat Only, No Iron: Participants on HD received roxadustat capsules at the applicable dose (up to a maximum roxadustat dose of 140, 200, and 300 milligrams [mg]) based on weight and hemoglobin (Hb) level, administered orally 3 times weekly (TIW) for 12 weeks.
- Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg: Participants on HD received roxadustat capsules at the applicable dose (up to a maximum roxadustat dose of 140, 200, and 300 mg) based on weight and Hb level, administered orally TIW with iron PO (ferrous fumarate or ferrous gluconate) at doses containing elemental iron between 50 and 195 mg daily (depending on the type of iron formulation available in their countries) for 12 weeks.
- Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg: Participants on HD received roxadustat capsules at the applicable dose (up to a maximum roxadustat dose of 140, 200, and 300 mg) based on weight and Hb level, administered orally TIW with approximately 60 mg IV iron (ferric gluconate complex in sucrose injection [for example, Ferrlecit®] or equivalent) once a week for 12 weeks.
- Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg: Participants on PD received roxadustat capsules at the applicable dose (up to a maximum roxadustat dose of 140, 200, and 300 mg) based on weight and Hb level, administered orally TIW with iron (ferrous fumarate or ferrous gluconate) PO at doses containing elemental iron between 50 and 195 mg daily (depending on the type of iron formulation available in their countries) for 12 weeks.
Period: Overall Study
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Started (Safety population: all participants who received any dose of study drug.) | 24 | 12 | 12 | 12
Efficacy Evaluable (EE) Population (All participants who received study treatment for 6 weeks or longer and had valid corresponding Hb measurements.) | 23 | 12 | 10 | 10
Completed | 21 | 12 | 10 | 10
Not Completed | 3 | 0 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Other than specified | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any dose of study drug.
Groups:
- Arm A + E (Participants on HD): Roxadustat Only, No Iron: Participants on HD received roxadustat capsules at the applicable dose (up to a maximum roxadustat dose of 140, 200, and 300 mg) based on weight and Hb level, administered orally TIW for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Total
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (17.7) | 46.8 (14.6) | 53.1 (12.6) | 51.4 (12.4) | 50.1 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 7 | 10 | 29
  Male | 15 | 9 | 5 | 2 | 31

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change From Baseline in Hb During Weeks 3-13
Description: Baseline Hb was defined as the mean of the last 3 central laboratory Hb values prior to the first dose administration. This outcome measure is derived from the maximum change from baseline during Weeks 3-13, without last observation carried forward (LOCF) imputation.
Time Frame: Baseline, Weeks 3-13
Population: EE population included participants who received study treatment for 6 weeks or longer and had valid corresponding Hb measurements.
Measure: Mean (Standard Error); unit: grams/deciliter (g/dL)
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
grams/deciliter (g/dL)
  Baseline | 8.1 (0.2) | 8.5 (0.3) | 8.4 (0.3) | 8.7 (0.2)
  Change at Weeks 3-13 | 2.8 (0.2) | 3.5 (0.5) | 3.5 (0.4) | 3.3 (0.2)
Statistical Analysis 1: Comparison: Arm A + E (Participants on HD): Roxadustat Only, No Iron vs Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg; Analysis of covariance (ANCOVA) model with treatment as a factor, baseline Hb and iron repletion status as covariates was used to compare treatments; Test type: Other; p = 0.0757, ANCOVA — Threshold for significance at 0.05 level
Statistical Analysis 2: Comparison: Arm A + E (Participants on HD): Roxadustat Only, No Iron vs Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg; ANCOVA model with treatment as a factor, baseline Hb and iron repletion status as covariates was used to compare treatments; Test type: Other; p = 0.0630, ANCOVA — Threshold for significance at 0.05 level
Statistical Analysis 3: Comparison: Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg vs Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.8653, ANCOVA — Threshold for significance at 0.05 level
Statistical Analysis 4: Comparison: Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg vs Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.8982, ANCOVA — Threshold for significance at 0.05 level

2. Secondary Outcome: Mean Change From Baseline in Hb During Weeks 2-5, 6-9, and 10-13
Description: Baseline Hb was defined as the mean of the last 3 central laboratory Hb values prior to the first dose administration.
Time Frame: Baseline, Weeks 2-5, 6-9, and 10-13
Population: EE population included participants who received study treatment for 6 weeks or longer and had valid corresponding Hb measurements. LOCF method was used to impute missing values.
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
g/dL
  Baseline | 8.1 (0.2) | 8.5 (0.3) | 8.4 (0.3) | 8.7 (0.2)
  Change at Weeks 2-5 | 1.1 (0.1) | 1.1 (0.2) | 1.0 (0.2) | 0.8 (0.3)
  Change at Weeks 6-9 | 2.0 (0.2) | 2.3 (0.4) | 2.0 (0.4) | 1.8 (0.4)
  Change at Weeks 10-13 | 2.1 (0.2) | 2.7 (0.5) | 3.0 (0.4) | 2.4 (0.2)

3. Secondary Outcome: Number of Participants Whose Maximum Hb Achieved During Treatment Was at Least 1.0 g/dL Increase From Baseline and Was ≥11.0 g/dL
Description: Baseline Hb was defined as the mean of the last 3 central laboratory Hb values prior to the first dose administration.
Time Frame: Week 3 to 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
Participants | 10 | 8 | 8 | 9

4. Secondary Outcome: Number of Participants Whose Maximum Hb Achieved During Treatment Was at Least 1.0 g/dL Increase From Baseline and Was ≥10.0 g/dL
Description: Baseline Hb was defined as the mean of the last 3 central laboratory Hb values prior to the first dose administration.
Time Frame: Week 3 to 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
Participants | 17 | 10 | 8 | 10

5. Secondary Outcome: Number of Participants With a Hb Response, Defined as an Increase in Hb by ≥1.0 g/dL From Baseline, by Weeks 5, 9, and 13
Description: Baseline Hb was defined as the mean of the last 3 central laboratory Hb values prior to the first dose administration.
Time Frame: Weeks 5, 9, and 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
Participants
  Week 5 | 21 | 9 | 7 | 7
  Week 9 | 22 | 10 | 9 | 9
  Week 13 | 22 | 11 | 10 | 10

6. Secondary Outcome: Number of Participants Who Achieved Maximum Hb During Weeks 3-13
Time Frame: Weeks 3-13
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
Participants
  <10 g/dL | 6 | 1 | 2 | 0
  10 to <11 g/dL | 7 | 3 | 0 | 1
  11 to 13 g/dL | 10 | 5 | 5 | 9
  >13 to 14 g/dL | 0 | 1 | 3 | 0
  >14 g/dL | 0 | 2 | 0 | 0

7. Secondary Outcome: Number of Participants With a Maximum Change From Baseline in Hb During Weeks 3-13
Description: Baseline Hb was defined as the mean of the last 3 central laboratory Hb values prior to the first dose administration. The number of participants who fall within the following categories of maximum change are reported: <1 g/dL, ≥1 g/dL, 1 to <2 g/dL, 2 to <3 g/dL, >3 to <4 g/dL, ≥4 g/dL.
Time Frame: Baseline, Weeks 3-13
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
Participants
  <1 g/dL | 1 | 1 | 0 | 0
  ≥1 g/dL | 22 | 11 | 10 | 10
  1 to <2 g/dL | 4 | 2 | 2 | 0
  2 to <3 g/dL | 9 | 2 | 0 | 5
  >3 to <4 g/dL | 7 | 2 | 4 | 3
  ≥4 g/dL | 2 | 5 | 4 | 2

8. Secondary Outcome: Median Time to Hb Response (Increase in Hb by ≥1.0 g/dL From Baseline)
Description: Baseline Hb was defined as the mean of the last 3 central laboratory Hb values prior to the first dose administration.
Time Frame: Baseline up to Week 13
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
weeks | 4.0 [3.0 to 4.0] | 4.0 [3.0 to 6.0] | 4.0 [3.0 to 6.0] | 4.0 [3.0 to 8.0]

9. Secondary Outcome: Weekly Dose at First Hb Response (Increase in Hb by ≥1.0 g/dL From Baseline)
Description: Baseline Hb was defined as the mean of the last 3 central laboratory Hb values prior to the first dose administration.
Time Frame: Baseline up to Week 13
Population: EE population included participants who received study treatment for 6 weeks or longer and had valid corresponding Hb measurements. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 22 | 11 | 10 | 10
mg/kg | 4.2 (0.5) | 4.2 (1.2) | 4.5 (1.4) | 4.3 (1.4)

10. Secondary Outcome: Number of Participants Requiring Dose Increase at Weeks 5 and 9
Description: Number of participants requiring dose increase due to any reasons is reported.
Time Frame: Weeks 5 and 9
Population: Safety population included all participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 24 | 12 | 12 | 12
Participants
  Week 5 | 2 | 3 | 2 | 4
  Week 9 | 8 | 5 | 3 | 5

11. Secondary Outcome: Number of Participants Requiring Dose Reduction or Dose Discontinuation Due to Excessive Erythropoiesis
Description: Number of participants requiring dose reduction or dose discontinuation due to excessive erythropoiesis is reported.
Time Frame: Weeks 5 and 9
Population: Safety population included all participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 24 | 12 | 12 | 12
Participants
  Dose reduced at Week 5 | 3 | 5 | 3 | 5
  Dose interrupted at Week 5 | 1 | 0 | 0 | 0
  Dose reduced at Week 9 | 1 | 0 | 3 | 0
  Dose interrupted at Week 9 | 1 | 0 | 0 | 1

12. Secondary Outcome: Change From Baseline in Ferritin at Week 13
Description: Baseline was defined as the average of the last 2 values prior to the first dose administration.
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Error); unit: micrograms/liter (µg/L)
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
micrograms/liter (µg/L)
  Baseline | 156.4 (12.9) | 162.5 (30.8) | 182.0 (27.4) | 137.4 (27.0)
  Change at Week 13 | -119.7 (12.2) | -51.1 (25.2) | -25.2 (33.5) | -65.1 (29.4)

13. Secondary Outcome: Change From Baseline in Transferrin Saturation (TSAT) at Week 13
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage of transferrin
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
percentage of transferrin
  Baseline | 18.8 (0.8) | 19.0 (1.0) | 18.1 (1.5) | 19.3 (1.8)
  Change at Week 13 | -7.4 (1.4) | 2.6 (2.5) | 0.7 (2.9) | -1.6 (2.6)

14. Secondary Outcome: Change From Baseline in Reticulocyte Hemoglobin Content at Week 13
Time Frame: Baseline, Week 13
Population: as for outcome 9
Measure: Mean (Standard Error); unit: picogram (pg)
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 21 | 10 | 10 | 10
picogram (pg)
  Baseline | 31.0 (0.3) | 31.6 (0.5) | 31.5 (0.5) | 30.4 (0.4)
  Change at Week 13 | -2.2 (0.7) | -1.9 (0.9) | -1.0 (0.6) | -0.2 (0.6)

15. Secondary Outcome: Number of Participants With Mean Hb Values 11.0-13.0 g/dL at Weeks 6-9 and 10-13
Time Frame: Weeks 6-9 and 10-13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
Participants
  Weeks 6-9 | 6 | 5 | 4 | 5
  Weeks 10-13 | 5 | 2 | 5 | 7

16. Secondary Outcome: Number of Participants With Mean Hb Values Within 11.0-13.0 g/dL During Weeks 10-13 Among Those With Maximum Hb ≥11.0 g/dL and Change of Hb ≥1 g/dL
Time Frame: Weeks 10-13
Population: EE population included participants who received study treatment for 6 weeks or longer and had valid corresponding Hb measurements. Here, 'Overall number of participants analyzed' signifies participants with maximum Hb ≥11 g/dL and change of Hb ≥1 g/dL during Weeks 10-13. LOCF method was used to impute missing values.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 10 | 8 | 8 | 9
Participants | 5 | 2 | 5 | 7

17. Secondary Outcome: Number of Participants With Mean Hb Values Within 10.0-13.0 g/dL During Weeks 10-13 Among Those With Maximum Hb ≥10.0 g/dL and Change of Hb ≥1 g/dL
Time Frame: Weeks 10-13
Population: EE population included participants who received study treatment for 6 weeks or longer and had valid corresponding Hb measurements. Here, 'Overall number of participants analyzed' signifies participants with maximum Hb ≥10 g/dL and change of Hb ≥1 g/dL during Weeks 10-13. LOCF method was used to impute missing values.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 17 | 10 | 8 | 10
Participants | 15 | 7 | 7 | 9

18. Secondary Outcome: Number of Participants With Mean Hb Values in Excess of 13.0 and 14.0 g/dL at Weeks 6-9 and 10-13
Time Frame: Weeks 6-9 and 10-13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
Participants
  Week 6-9 | 0 | 0 | 0 | 0
  Week 10-13 | 0 | 1 | 1 | 0

19. Secondary Outcome: Number of Participants With Mean Hb Values <10.0 g/dL at Weeks 6-9 and 10-13
Time Frame: Weeks 6-9 and 10-13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
Participants
  Week 6-9 | 10 | 4 | 2 | 3
  Week 10-13 | 8 | 3 | 2 | 1

20. Secondary Outcome: Number of Participants Requiring Rescue Treatment With an Erythropoiesis-Stimulating Agent (ESA), Red Blood Cells (RBC) Transfusion, or IV Iron (Excluding Arm C)
Description: Number of participants requiring rescue treatment with an ESA, RBC transfusion, or IV Iron (Excluding Arm C) was reported.
Time Frame: Baseline up to Week 13
Population: Safety population included all participants who received any dose of study drug. Here 'Number analyzed' signifies participants evaluable for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 24 | 12 | 12 | 12
Participants
  Blood transfusion for severe anemia | 0 | 0 | 1 | 0
  Blood transfusion for gastrointestinal bleeding | 1 | 0 | 0 | 0
  IV iron for acute iron deficiency: number analyzed (Participants) | 24 | 12 | 0 | 12
  IV iron for acute iron deficiency | 1 | 0 |  | 0
  IV iron for a treatment-emergent adverse event (TEAE) of thrombocytosis: number analyzed (Participants) | 24 | 12 | 0 | 12
  IV iron for a treatment-emergent adverse event (TEAE) of thrombocytosis | 1 | 0 |  | 0

21. Secondary Outcome: Number of Participants Requiring Therapeutic Phlebotomy
Description: Number of participants who required therapeutic phlebotomy due to TEAE of abnormal erythropoiesis is reported.
Time Frame: Baseline up to Week 13
Population: Safety population included all participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 24 | 12 | 12 | 12
Participants | 0 | 1 | 0 | 0

22. Secondary Outcome: Number of Participants Withdrawn From the Study Due to Inadequate Efficacy
Description: Number of participants withdrawn from the study due to inadequate efficacy is reported.
Time Frame: Baseline up to Week 16
Population: Safety population included all participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 24 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline in Short Form 36 (SF-36) Version 2 Physical Functioning Subscore and Vitality Subscore at Weeks 9 and 13
Description: The SF-36 V2 consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems, role limitations due to emotional problems, general health perceptions, mental health, social function, and vitality. The physical functioning subscore and vitality subscore are reported. The scores ranged from 0 (worst) to 100 (Best). Higher score indicated a better health state. Baseline is defined as the last non-missing value prior to the first dose administration.
Time Frame: Baseline, Weeks 9 and 13
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
units on a scale
  Physical functioning subscore: Baseline | 38.8 (2.3) | 40.7 (3.2) | 41.2 (3.4) | 40.8 (1.8)
  Physical functioning subscore: Change at Week 9 | 4.8 (1.6) | 1.6 (2.5) | 1.5 (2.5) | 3.4 (1.2)
  Physical functioning subscore: Change at Week 13 | 5.2 (1.8) | 1.8 (2.1) | 4.8 (1.8) | 2.3 (1.3)
  Vitality subscore: Baseline | 46.3 (2.2) | 48.2 (4.1) | 49.0 (3.5) | 46.8 (3.6)
  Vitality subscore: Change at Week 9 | 2.9 (1.8) | -1.0 (4.0) | 3.4 (2.8) | 5.9 (3.0)
  Vitality subscore: Change at Week 13 | 3.9 (1.7) | 1.6 (3.7) | 3.1 (2.3) | 6.2 (1.6)

24. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Anemia (FACT-An) Total Score at Weeks 9 and 13
Description: FACT-An is composed of 27 core items which assess participant's function in 4 domains and 20 anemia-related items, grouped into 5 subscales as follows: Physical well-being (PWB): 7 items; Social/family well-being (SWB): 7 items; Emotional well-being (EWB): 6 items; Functional well-being (FWB): 7 items; and Anemia: 20 items. All FACT-An items were rated as: 0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much. Each subscale score was the sum of scores for the items in the subscale. The FACT-An total score was the sum of all 5 subscale scores, ranging from 0 (worst) - 188 (best). Higher scores represented better quality of life. Baseline is defined as the last non-missing value prior to the first dose administration.
Time Frame: Baseline, Weeks 9 and 13
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 23 | 12 | 10 | 10
units on a scale
  Baseline | 123.5 (6.8) | 118.9 (10.9) | 128.8 (11.3) | 122.8 (7.9)
  Change at Week 9 | 8.2 (4.5) | 4.0 (7.2) | 1.9 (9.8) | 12.8 (6.9)
  Change at Week 13 | 7.3 (4.3) | 5.9 (6.9) | 5.1 (8.9) | 12.9 (7.4)

25. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Tests
Description: Criteria for the potential clinical significance included: bilirubin (µmol/L) >1.5 * upper limit of normal (ULN), potassium (mmol/L) >1.2 * ULN, neutrophils (*10^9/L) ≤1, protein (g/L) >1.1 * ULN, leukocytes (*10^9/L) ≤2.5 or ≥15.
Time Frame: Baseline up to Week 16
Population: Safety population included all participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 24 | 12 | 12 | 12
Participants
  Bilirubin | 1 | 0 | 0 | 0
  Potassium | 2 | 1 | 0 | 1
  Neutrophils | 0 | 1 | 1 | 0
  Protein | 1 | 0 | 0 | 0
  Leukocytes | 1 | 0 | 1 | 0

26. Secondary Outcome: Number of Participants With TEAEs
Description: An adverse event (AE) was any untoward medical event in a participant who received study drug whether or not the event is considered drug related. TEAEs were defined as any event that either began or worsened after the first administration of study drug and within 28 days of the last dose. A summary of other nonserious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 16
Population: Safety population included all participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Number analyzed (Participants) | 24 | 12 | 12 | 12
Participants | 16 | 6 | 3 | 5

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Description: Safety population included all participants who received any dose of study drug. Non-serious adverse events are reported in the section labeled "Other Adverse Events".
Arm/Group | Arm A + E (Participants on HD): Roxadustat Only, No Iron | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg
Serious Adverse Events (participants affected / at risk) | 3/24 | 1/12 | 0/12 | 3/12
Other Adverse Events (participants affected / at risk) | 6/24 | 4/12 | 0/12 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A + E (Participants on HD): Roxadustat Only, No Iron (N=24) | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg (N=12) | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg (N=12) | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg (N=12)
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A + E (Participants on HD): Roxadustat Only, No Iron (N=24) | Arm B (Participants on HD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg (N=12) | Arm C (Participants on HD): IV Iron (Ferric Gluconate Complex in Sucrose or Equivalent) 60 mg (N=12) | Arm D (Participants on PD): PO Iron (Ferrous Fumarate or Ferrous Gluconate) Between 50 and 195 mg (N=12)
Transferrin saturation decreased (Investigations) | 3 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 3 | 0 | 2
Phlebitis (Vascular disorders) | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes